CLINICAL TRIAL: NCT02822365
Title: Calibrated Methods for Quantitative PET/CT Imaging Phase II
Brief Title: Pocket Phantom Tool in Improving Accuracy of Quantitative PET/CT Imaging of Patients With Solid Tumors
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9592; NCI-2016-00747 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9592 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); R42CA167907 (NIH)
Record Dates: First submitted 2016-06-22; First posted 2016-07-04 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Adult Solid Neoplasm
MeSH Terms: interventions — Phantoms, Imaging; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic (PET/CT): Patients undergo a PET/CT scan as part of their standard clinical care. While still positioned for the clinical scan, patients undergo additional research PET/CT scans in a smaller region over 10 minutes with the pocket phantom placed nearby and a low-dose single bed position CTAC.
  Interventions: Procedure: Computed Tomography; Device: Imaging Phantoms; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scan as clinically indicated (Note: CT is for attenuation correction and not for diagnostic purposes).
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Device: Imaging Phantoms — Undergo limited field of view PET scan with the Pocket Phantom placed nearby to assist in scanner calibration. No additional PET tracer will be used.
  Other Names: Phantoms
Procedure: Positron Emission Tomography — Undergo PET/CT scan as clinically indicated.
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot study tests the pocket phantom tool in improving the accuracy of quantitative positron emission tomography/computed tomography (PET/CT) imaging of patients with solid tumors. The pocket phantom tool may help test the accuracy of the PET/CT scanner and indicate whether adjustments need to be made to get consistent information.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Optimize the pocket phantom source design and the bias estimation algorithm: determine the tolerances and variations in the source sphere geometry and radioactive filing process; evaluate the need for higher-activity sources in the presence of increased attenuation (i.e. thicker patients); optimize CT contrast levels for source boundary detection and localization from CT images; evaluate the robustness for use with different scanner parameters (e.g. CT slice thicknesses); modify bias estimation algorithm as needed to take into account changes.

II. Develop automated and robust ID pocket phantom processing and web-based software as a service (SAS) analysis tools: automate initial identification of approximate location of the pocket phantom; add automated DICOM analysis for web-based SAS analysis tools for imaging sites.

III. Conduct phantom studies at multiple imaging centers to evaluate the performance with different imaging protocols, scanners, and reconstruction methods. Also test at multiple time points over 6-9 months to assess longitudinal stability.

IV. Conduct a comparative study with patients (at University of Washington [UW]) at multiple time points over 6-12 months to evaluate the performance of the pocket phantom in oncology patient imaging compared with current clinical practice.

OUTLINE:

Patients undergo a PET/CT scan as part of their standard clinical care. While still positioned for the clinical scan, patients undergo additional research PET/CT scans in a smaller region over 10 minutes with the pocket phantom placed nearby and a low-dose single bed position CT scan for attenuation correction (CTAC).

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving clinically indicated PET/CT scan
* Patient has a known solid tumor
* Patient provides consent
* Patient can tolerate additional time in scanner (i.e. not claustrophobic)

Exclusion Criteria:

* Patient is pregnant
* Patient cannot or does not provide consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors receiving clinically indicated PET/CT scans.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Difference in measured versus known quantitative values of the pocket phantom | At day 1 (All data will be collected during the clinically scheduled appointment. Analysis will follow typical image reconstruction times.)
  Compare measured activity of the pocket phantom (as measured by a PET/CT scanner) to the known values of the pocket phantom (as calculated based on half-life activity of known source) to determine accuracy and precision of scanner calibration. This will be used to validate quantitative clinical measurements, like SUV (standardized uptake values), of known solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kinahan, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States